CLINICAL TRIAL: NCT05575180
Title: Effect of Acetazolamide and Methazolamide on Hypoxic Exercise Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Wilderness Medical Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 43720
Record Dates: First submitted 2022-09-08; First posted 2022-10-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-09

CONDITIONS: High Altitude Effects
Keywords: exercise
MeSH Terms: conditions — Altitude Sickness; Motor Activity | interventions — Acetazolamide; Methazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methazolamide (Experimental): Drug: Methazolamide Dose: 100 mg b.i.d Duration: 2 days prior to testing + 1 hr prior to testing start Form: Oral
  Interventions: Drug: Methazolamide Pill
- Acetazolamide (Active Comparator): Drug: Acetazolamide Dose: 250 mg t.i.d Duration: 2 days prior to testing + 1 hr prior to testing start Form: Oral
  Interventions: Drug: Acetazolamide 250Mg Tab
- Placebo (Placebo Comparator): Drug: Placebo (microcrystalline cellulose) Dose: 250 mg t.i.d Duration: 2 days prior to testing + 1 hr prior to testing start Form: Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide 250Mg Tab — Oral acetazolamide
  Arms: Acetazolamide
Drug: Methazolamide Pill — Oral Methazolamide
  Arms: Methazolamide
Drug: Placebo — Oral placebo
  Arms: Placebo

SUMMARY:
A single-centered randomized doubled blinded placebo-controlled cross-over trial comparing two the effect of two carbonic anhydrase inhibitors on exercise performance in acute hypoxia. Participants will be young (under 40 years of age), healthy males and females who are regularly physically active.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided
* Between ages of 18-40 years old
* In good general health as evidences by medical history
* Perform at least 150 mins of aerobic exercise per week, and engage in physical activity >2 days a week
* Completed in an endurance event in the last 12 months
* Ability to take oral medication, and be willing to adhere to the drug regimen
* Be willing to have blood samples taken

Exclusion Criteria:

* Weigh 49kg or less, or are Obese (BMI >30 kg/m2)
* Presence of chronic health condition (s), being investigated and/or taking prescription medications for the following disorders:

  1. Cardiovascular - e.g., hypertension
  2. Metabolic - e.g., type 1 or 2 diabetes
  3. Respiratory - e.g., chronic obstructive pulmonary disease, asthma
  4. Digestive - e.g., ulcerative colitis
  5. Arthritis
  6. Cancer
* Presence of any disorder or condition listed in the health screening questionnaire (see section 12.1)
* Current use of Lonafarnib, Methenamine, Topamax, or steroids/corticosteroids
* Known allergic reactions/hypersensitivity to carbonic anhydrase inhibitors or sulfonamides
* Presence of bleeding or clotting disorders
* Current smoker or cannabis user
* Pregnant, suspect to be pregnant, currently planning a pregnancy, or nursing
* Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Time to complete a 5 km time trial after each experimental day (Days 3-5) | The time to complete the 5 km time trial is measured after each time trial. The investigators will be blinded until all participants have completed each trial
  Primary endpoint is the time to complete a 5 km exercise task in the three arms of the trial (acetazolamide, methazolamide, placebo)

SECONDARY OUTCOMES:
Expired Minute Ventilation | The average minute ventilation for each time trial km (1-5) for each arm will be determined. The investigators will be blinded until all participants have completed each trial
  The secondary endpoint expired minute ventilation will be measured using a flow meter (pneumotach) which measure flow and allows for the calculation of ventilation. The value is expressed in liters per min and measured continuously
Oxyhemoglobin saturation | The average oxyhemoglobin saturation for each time trial km (1-5) for each arm will be determined. The investigators will be blinded until all participants have completed each trial
  The secondary endpoint oxyhemoglobin saturation will be measured using a pulse oximeter which measure the fraction of hemoglobin bound to oxygen. The value is expressed as a percent and measured continuously

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada